CLINICAL TRIAL: NCT03948724
Title: Randomized Controlled Trial Evaluating the Impact of Therapeutic Patient Education on the Toxicity of Immune Checkpoint Inhibitors in Oncology
Brief Title: Impact of Therapeutic Patient Education on the Toxicity of Immune Checkpoint Inhibitors in Oncology
Acronym: EDHITO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICO-2019-02
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Therapeutic Patient Education; Immune Checkpoint Inhibitors; Melanoma; Advanced Non-small Cell Lung Cancer; Renal Cell Carcinoma; Head and Neck Cancer; Immune-related Adverse Event
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic patient education (Experimental): Patient will receive 5 therapeutic education sessions.
  Interventions: Behavioral: Therapeutic education program
- Standard Care (Active Comparator): Patient will receive usual informations
  Interventions: Behavioral: Usual Information

INTERVENTIONS:
Behavioral: Therapeutic education program — Patient will have 5 educational therapy workshops. The first educational therapy workshops will be realized at cycle 1 and the last one within 25 weeks after starting treatment
  Arms: Therapeutic patient education
Behavioral: Usual Information — Patient receive usual informations
  Arms: Standard Care

SUMMARY:
The aim of this therapeutic education program is to reduce the apparition of immune-related Adverse Event with patients treated with ICI

DETAILED DESCRIPTION:
This study aims to highlight the impact of Patient Therapeutic Education (TPE) in oncology. TPE is an integral part of the care pathway for patients with a chronic pathology such as diabetes, asthma, chronic obstructive pulmonary disease, cardiovascular diseases requiring anticoagulants, haemophilia, renal failure, HIV infection, autoimmune diseases etc.... front of therapeutic progress, many cancers are now taken for a chronic disease.

In oncology, TPE starts to grow. Indeed, TPE makes the patient more autonomous, which could reduce the occurrence and / or aggravation of some toxicities, improve the quality of life, the effectiveness of treatment and optimize health costs. Therefore, it is important to develop programme of therapeutic education in oncology.

The toxicity of ICI is unusual and sometimes lethal. This toxicity must be recognized and managed quickly to maintain a satisfactory dose-intensity. TPE finds its place by raising awareness among patient to the occurrence of these toxicities.

This randomized TPE versus standard care study project will assess the contribution of education in the management of severe toxicities. The investigators believe that changes in patient behaviour will reduce the number of toxicities ≥3 in the TPE arm.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Melanoma, Non-Small Cell Bronchial Cancer, renal cell carcinoma, Ca carcinomas of the upper airways to be treated with ICI
* Patient who has never received treatment by ICI
* Informed patient who signed his consent
* Age > or = 18 years
* Social insurance

Exclusion Criteria:

* Patient receiving corticosteroid or immunosuppressant 14 days before inclusion
* Immunocompromised patient
* Uncontrolled brain metastases
* Refusal to participate, patient protected by guardianship
* Patient unable to understand the study or unable to follow the education sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Comparison of the number of patients with at least one grade ≥ 3 immune-related Adverse Event (irAE) toxicity for 25 weeks after initiation of ICI treatment between both arm | 36 months
  Measure of the number of patients with at least one immune-related Adverse Event (irAE) grade ≥ 3 (CTCAE v5.0) for 25 weeks following the beginning of ICI treatment.

SECONDARY OUTCOMES:
Characterize the toxicity of Immune Checkpoint Inhibitors (ICI) | 36 months
  Description of immune-related Adverse Event of grade> 2
Quantification of ICI treatment received | 36 months
  Description of each cycle of ICI
Measuring the level of knowledge of patients related to the disease, the treatment and its side effects | 36 months
  Measuring the level of knowledge of patients with a specific questionnaire
Patients' quality of life assessment: Hospital Anxiety and Depression Scale | 36 months
  quality of life evaluated with the Hospital Anxiety and Depression Scale
Patients' quality of life assessment: questionnaire-C30 | 36 months
  quality of life evaluated with the Quality-of-life questionnaire-C30

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Beaumont, Principal Investigator — INSTITUT DE CANCEROLOGIE DE L'OUEST
Locations (9):
- France (9):
  - Chu Angers, Angers
  - Institut de Cancerologie de L'Ouest, Angers
  - Centre Francois Baclesse, Caen
  - Centre D'Oncologie Et de Radiotherapie 37, Chambray-lès-Tours
  - Chd Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No